CLINICAL TRIAL: NCT06806332
Title: Glaucoma Drop Aids Part 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston Medical Center Patient Safety Grant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45629
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma; Intraocular Pressure
Keywords: Eye drop aid; Nanodropper
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Drop aid used then no drop aid (Experimental): Participants randomized into this group will be assigned to use the Nanodropper over the first 4-6 weeks, and then no drop aid device over the next 4-6 weeks.
  Interventions: Device: Nanodropper
- No drop aid then drop aid (Experimental): Participants randomized into this group will be assigned to use no drop aid over the first 4-6 weeks, and then to use the Nanodropper over the next 4-6 weeks.
  Interventions: Device: Nanodropper

INTERVENTIONS:
Device: Nanodropper — The Nanodropper is the only FDA-listed, volume-reducing adaptor for eyedrop bottles. By twisting the Nanodropper onto a compatible bottle, the drop-size can be reduced by over 60%. Smaller drops have been shown to reduce waste, cost, and side effects.
  Other Names: Drop aid

SUMMARY:
Glaucoma medications are vital to disease management and prevention of further loss of vision as over time glaucoma will lead to irreversible blindness. The average size of a glaucoma medication bottle is around 10cc and these medications when used 2-3 times daily are expected to last patients an entire month. The investigators found that at Boston Medical Center (BMC) a majority of Yawkey Eye Clinic patients are unable to deliver the drops into their eyes due to poor vision or difficulty squeezing drop bottles. These patients also often deliver more than a necessary amount leading to premature completion of the bottle. However, because the cost benefit ratio of these drop aids is unclear, they are not routinely offered to the patients. Although the efficacy of these drop aids has not been well studied, if effective, the cost of these drop aids would more than pay themselves by improving medication compliance and visual function of the patients. This study aims to determine the efficacy of the Nanodropper in the BMC Yawkey Eye Clinic patient population.

DETAILED DESCRIPTION:
A randomized, crossover study design will be used to determine the efficacy of the Nanodropper in the BMC Yawkey Eye Clinic patient population. All participants will receive the Nanodropper, but will be randomly assigned to study groups defined by the order in which they use the Nanodropper. The first group will be assigned to use the drop aid device over the first 4-6 weeks, and then no drop aid device over the next 4-6 weeks. The second group will be assigned to use no drop aid device over the first 4-6 weeks, and then the drop aid device over the next 4-6 weeks. Therefore, each participant will undergo two study periods (using the drop aid and not using the drop aid).

Prior to use of the Nanodropper, participants will be instructed on how to use the drop aid by a member of the research team and a preintervention intraocular pressure check will be performed using an applanator which is part of the patient's standard of care. Intraocular pressure is the only adjustable risk factor for glaucoma; thus, glaucoma treatments slow progression of glaucoma by reducing intraocular pressure.

After 3 weeks and after at least 6 weeks per study period, participants will complete a satisfaction survey for the drop aid treatment group or control group. The 3 week satisfaction survey will take place over the phone. As part of routine eye care, participants will need to return to the clinic at least 6 week after enrollment. During this visit, a satisfaction survey will be completed, the participant's study diary will be collected, and routine intraocular pressure checks will be documented. If the participant does not complete the home study diary or forgets to bring it in to their appointment, a member of the study team will help them fill it out at a follow-up clinic appointment. The duration of participation for each subject will be 8-12 weeks.

The efficacy of the Nanodropper will be compared to the control and measured with any changes in intraocular pressure readings, length of time to medication completion, and patient satisfaction according to the surveys.

ELIGIBILITY:
Inclusion Criteria:

* Currently on the same topical ophthalmic medications for treatment of glaucoma for a minimum of two months
* Patient of Boston University Eye Associates

Exclusion Criteria:

* Changed glaucoma medications within the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Completion of topical ophthalmic drug bottle | 12 weeks
  This outcome will be measured in days by the patient from when a bottle is started until all the medication has been used.
Satisfaction with dispensing opthalmic medication | 12 weeks
  An investigator developed survey completed by participants will be used to assess participants' satisfaction of eye drops with and without the drop aid.

SECONDARY OUTCOMES:
Change in intraocular pressure with drop aid | before starting the drop aid, after 6 weeks of using the drop aid
  An applanator will be used to measure the intraocular pressure during standard of care appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Manishi Desai, MD, Principal Investigator — BostonMedical Center, Ophthalmology
Locations (1):
- Yawkey Eye Clinic, Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No